CLINICAL TRIAL: NCT02657811
Title: Time-Lapse Incubation for Embryo Culture - The Impact of Morphokinetics and Environmental Stability on Reproductive Outcomes
Brief Title: Time-Lapse Incubation for Embryo Culture - Morphokinetics and Environmental Stability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Ruthie Ronn, Dr. Ruth Ronn, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0169-15-SZMC
Record Dates: First submitted 2016-01-05; First posted 2016-01-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Infertility; Genetic Diseases
Keywords: Time-Lapse Imaging; Embryo Culture Techniques; Fertilization in Vitro; Embryology; Assisted Reproductive Techniques; Infertility; Preimplantation diagnosis
MeSH Terms: conditions — Infertility; Genetic Diseases, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bench Incubation (Active Comparator): These embryos will be randomized to the bench incubator.
  Interventions: Device: Miri, Benchtop Multi-room incubator
- Time Lapse Incubation (Active Comparator): These embryos will be randomized to the Time Lapse Incubator.
  Interventions: Device: Miri TL, Time-Lapse incubator
- Time Lapse Incubation - Modified (Active Comparator): These embryos will be randomized to the bench incubator.
  Interventions: Device: Miri TL, Time-Lapse incubator

INTERVENTIONS:
Device: Miri, Benchtop Multi-room incubator — Bench Incubation - Morphologic Assessment These embryos will undergo multiple evaluations using light microscopy and traditional morphologic assessment.
  Arms: Bench Incubation
Device: Miri TL, Time-Lapse incubator — Time Lapse Incubation - Morphologic/Morphokinetic Assessment These embryos will remain in the TLI and undergo both morphologic and morphokinetic evaluation and grading according to a hierarchical multivariable model. They will not be removed from incubation for the duration of culture.
  Arms: Time Lapse Incubation
Device: Miri TL, Time-Lapse incubator — Time Lapse Incubation - Morphologic Assessment These embryos will remain in the TLI and undergo only traditional morphologic assessment according to accepted criteria with no additional imaging. They will also not be removed from incubation for the duration of culture. The time points and evaluated parameters will be identical to those in arm 1 of the study.
  Arms: Time Lapse Incubation - Modified

SUMMARY:
Embryo culture and selection has been a continuous challenge in evolution since the birth of In Vitro Fertilization (IVF). Traditionally, embryo quality and its presumed suitability for transfer were assessed based on morphologic features. However, the consensus as to the optimal time points for embryo assessment and as to 'preferable' characteristics have been challenging. Alongside this has been the challenge of achieving balance between multiple points of assessment, yet stabilizing the embryo environment for growth. In standard incubation, each new morphological assessment of embryos in culture theoretically creates an additional disruption to culture.

Most recently, time-lapse incubators (TLI) have been introduced as a novel embryo culture system attempting to limit culture disturbances. These incubators have been integrated with digital imaging, allowing for a substantial limitation in embryo handling and environmental disturbances. They have also introduced new morphokinetic parameters to embryo assessment and to optimizing selection of embryos. Thus far, a limited number of studies have examined the clinical outcomes and value of time lapse monitoring systems versus the more ubiquitous incubators (e.g. multichamber) for reproductive outcomes. In particular, the isolated value of morphokinetics in embryo assessment and of this new stable culture environment in TLI are still in question.

The objectives of this study are to prospectively assess and compare fertility outcomes when embryos are cultured in the TLI system versus more traditional bench incubators (BI). We will specifically assess the added value of the closed and isolated TLI compared to BI on reproductive outcomes, as well as the value of morphokinetic grading in IVF.

DETAILED DESCRIPTION:
Research Objectives:

We are now reaching a new age with an opportunity to advance to theoretically better culture environments and improvements on measures of embryo assessment.

The objectives of this research study will be to evaluate and compare the reproductive outcomes in isolating one of two new interventions introduced by the Time-Lapse Incubator (TLI) system. The first will be an assessment of the TLI environment compared to the standard Bench Incubator (BI) environment. The second will be an assessment of the added morphokinetic grading of embryos compared to the traditional morphologic grading alone.

Although the primary objective of this study will focus on clinical pregnancy rates and fresh embryo transfers, further research using embryos frozen from this study will be conducted to also evaluate cumulative pregnancy rates per oocyte pick-up (OPU) cycle in the future.

Methods The current study will be a prospective randomized and double-blinded study using three patient arms. The first arm will include patients randomized to embryo culture in a tri-gas bench incubator (Miri, Benchtop Multi-room incubator). These embryos will undergo multiple evaluations using light microscopy and traditional morphologic assessment according to accepted criteria. The second arm will include patients randomized to embryo culture in a time-lapse incubator (Miri TL, Time-Lapse Incubator). These embryos will remain in the TLI and undergo both morphologic and morphokinetic evaluation and grading according to a multivariable scoring model. They will not be removed from incubation for the duration of culture. The third arm will include patients also randomized to embryo culture in a time-lapse incubator (Miri TL, Time-Lapse Incubator). These embryos will remain in the TLI and undergo only traditional morphologic assessment according to accepted criteria with no additional imaging. They will also not be removed from incubation for the duration of culture. The time points and evaluated parameters will be identical to those in arm 1 of the study.

Patients will be assessed for suitability, inclusion and exclusion criteria by the physician and nursing team prior to initiation of an IVF/ICSI cycle at our centre. Once the patient is deemed eligible, a member of the care team will discuss details of the study with the patient.

Approved study subjects will undergo standard controlled ovarian hyperstimulation (COH). Protocols and their corresponding medications will be decided upon at the discretion of the treating physician. These may include long gonadotropin-releasing hormone (GnRH) agonist protocol and GnRH antagonist protocol. Follicular aspiration will be performed in the IVF unit via transvaginal needle aspiration. Endometrial preparation and luteal phase support will be recommended as per our departmental protocol. The number of embryos for transfer will be defined prior to cycle initiation, according to The Israel Society of Obstetrics & Gynecology.

Patient randomization will occur after Human Chorionic Gonadotropin (hCG) administration has already been ensured, prior to Intracytoplasmic Sperm Injection (ICSI). The randomization procedure will be accomplished using computer-generated randomization.

After follicular aspiration and transfer to the laboratory, the follicular fluid will be examined for presence of oocytes. Oocytes will then be scored for maturity and any morphologically abnormal features. ICSI will then be performed using fresh sperm from the corresponding partner.

Embryos will then be placed in culture media. The embryos within culture media will then be placed in either the Miri Benchtop or Miri Timelapse incubator according to their corresponding group of randomization. Note that the environment of the Miri benchtop and Miri TL incubators will be considered identical. oxygen concentration and carbon dioxide concentrations set at 5% and 5.5% respectively.

Embryos in arm 1 of the study (Miri Benchtop incubator) will be morphologically assessed by light microscopy at pre-defined time points and according to accepted criteria by one of the trained laboratory embryologists. The time points for evaluation will be at 16 - 20 hours post-ICSI (for normal fertilization), at 44 - 48 hours (day 2) post-ICSI, and then at 64 - 72 hours (day 3) post-ICSI. Evaluated parameters will include cell number, cell size, cell symmetry, and percent fragmentation. Any gross abnormalities will be noted. Embryos will then be graded on day 3 according to these evaluated parameters and transferred according to preferential grading. If embryo transfer has been predetermined for day 5, additional assessment will take place at approximately 116 hours.

Embryos in arm 2 of the study (Miri TL incubator) will be morphologically and morphokinetically assessed by the same laboratory embryologists using digital images generated by the incubator's integrated time-lapse imaging system. Assessment and scoring will be performed as per our scoring classification system. Morphological screening of embryos will initially be performed in order to discard or exclude those clearly not viable for transfer. Morphokinetic parameters will then be used in order to rank remaining embryos score categories from a maximum of 4.0 to a minimum of -2.0, in order of hypothesized decreasing implantation potential.

Embryos in arm 3 of the study (Miri TL incubator) will be morphologically assessed by the embryologists using digital images generated by the incubator's integrated time-lapse imaging system. As noted above, the time points and evaluated parameters will be identical to those in arm 1 of the study. Decisions on embryos for transfer will also be identical.

For each patient, embryos will be selected for transfer based on their morphologic scoring alone (Arm 1 and 3) or by the morphokinetic decision tree scoring (Arm 2). The number of embryos for transfer will have been pre-determined (as noted above).

Those embryos not selected and deemed appropriate for future transfer will undergo cryopreservation by vitrification.

Blinding of the current study will be ensured at multiple points. The gynecologists performing oocyte retrieval and embryo transfer will be blinded to the predefined and randomized patient group. Patients will be unaware of their group of randomization. Statisticians will also be blinded to the group of randomization in calculating pregnancy outcomes. It will unfortunately not be possible to ensure blinding of those embryologists performing the morphologic and morphokinetic assessments.

Sample Size calculation:

The pregnancy rate in our IVF Unit in the sub-group of patients with demographic and clinical characteristics similar to those included in the study, is about 40%. Assuming that in the TLI group pregnancy rate will increase by 10%, the sample size required per group is 124 patients per arm, with an alpha risk of 5% and a power of 80%.

Statistics:

The statistical analysis will be done by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring assisted reproductive technologies for one or more of the following reasons:

  * Male factor infertility
  * Unexplained infertility
  * Mechanical factor infertility
  * Ovulatory infertility
* Patients undergoing fertility treatment at Shaare Zedek Medical Centre alone.
* Patients attempting pregnancy with autologous gametes.
* Patients receiving embryo transfers according to the Israel Society of Obstetrics and Gynecology guideline on number of embryos for transfer during in vitro fertilization.
* Patients undergoing their first or second ICSI cycle (cumulative to all other institutions involved in prior treatment) since their previous pregnancy.
* BMI criteria: >18 and <30 kg/m2

Exclusion Criteria:

* An infertility diagnosis that includes the following:

  * Severe male factor infertility requiring testicular aspiration, testicular biopsy for sperm retrieval, or less than 1000 sperm per ejaculate.
  * Untreated hydrosalpinx
  * Persistently thin endometrial lining or endometrial factor
  * Severe Endometriosis
  * Low ovarian reserve (≤8 antral follicle count (AFC) follicles measuring 2 to 10 mm in diameter on day 2-4 of menstrual cycle, or day 3 follicle stimulating hormone (FSH) ≥10 milli-International unit (mIU) /mL)
  * High risk for Ovarian Hyperstimulation Syndrome (Estradiol level >13 000 pmol/L or >20 follicles ≥16 mm diameter during controlled ovarian hyper stimulation, ≥20 oocytes collected).
* Patients obtaining GnRH agonist for final follicular maturation
* Patients requiring preimplantation genetic diagnosis (PGD)
* Patients who require freezing of all oocytes or embryos
* More than 2 previous cycles of IVF since previous pregnancy
* Current smokers

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 372 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks gestation
  The number of women with a viable pregnancy (including gestational sac and fetal heart beat) at 12 weeks gestation divided by the number of women having an embryo transfer.

SECONDARY OUTCOMES:
Embryo morphology - Number of pronuclei present following fertilization | Day 1 post-fertilization
  Number of pronuclei present in the embryo 1 day following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - Number of cells present | Day 2 and Day 3 post-fertilization
  Number of cells present in the embryo 2 and 3 days following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - % fragmentation | Day 2 and Day 3 post-fertilization
  Percent fragmentation in the embryo 2 and 3 days following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - Presence of multi nucleation | Day 2 post-fertilization
  Presence of multi-nucleation in the embryo on day 2 following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - Symmetry | Day 2 and Day 3 post-fertilization
  Symmetry in the embryo 2 and 3 days following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - Stage of development at day 5 | Day 5 post-fertilization
  Stage of development in the embryo 5 days following fertilization. Characterized as: Early blastocyst, Blastocyst, Expanded, Hatched/Hatching, or other. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - Inner Cell Mass (ICM) grade | Day 5 post-fertilization
  ICM grade in the embryo 5 days following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphology - Trophectoderm grade | Day 5 post-fertilization
  Trophectoderm grade in the embryo 5 days following fertilization. Morphologic assessment parameter used to grade embryo quality.
Embryo morphokinetics - Abrupt division | Day 0 to Day 3 post-fertilization
  Presence or absence of abrupt division of the embryo from one to three or more cells: a morphokinetic assessment parameter used to grade embryo quality.
Embryo morphokinetics - Time of cleavage to five-blastomere embryo | Day 0 to Day 3 post-fertilization
  Presence or absence of optimal time range for cleavage to five-blastomere embryo (48.8-56.6 hours): a morphokinetic assessment parameter used to grade embryo quality.
Embryo morphokinetics - Time from two to four-blastomere embryo | Day 1 to Day 3 post-fertilization
  Presence or absence of optimal time duration of division from 2 to 3 cells and subsequent division to 4 cells (0-0.76 hours): a morphokinetic assessment parameter used to grade embryo quality.
Embryo morphokinetics - Time from two to three-blastomere embryo | Day 1 to Day 3 post-fertilization
  Presence or absence of optimal time duration of division from two-cell to three-cell embryo (0-11.9 hours): a morphokinetic assessment parameter used to grade embryo quality.
Oocyte characteristics - Polar body presence | Oocyte retrieval until fertilization - less than 1 day
  Polar body presence of oocyte on day of oocyte retrieval
Biochemical pregnancy rate | 14 days after embryo transfer
  The number of women with a positive β-hCG approximately 14 days after embryo transfer divided by the number of women having an embryo transfer.
Cumulative ongoing pregnancy rate | One year from oocyte pickup
  Cumulative number of women with a viable pregnancy at 12 weeks (where pregnancy was obtained with fresh and vitrified embryos from the same ovarian stimulation cycle) divided by the number of women having undergone an oocyte pickup cycle.
Live birth rate | One year and forty weeks
  The percentage of all Oocyte Pick Up (OPU) cycles that lead to live birth Approximate time frame will be time of one ovarian stimulation cycle plus term pregnancy
Spontaneous abortion rate | First 20 weeks of gestation
  Loss of an embryo or fetus prior to 20 weeks gestation or weighing less than 500 grams.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Ronn, M.D. C.M., Principal Investigator — Shaare Zedek Medical Center; Talia Eldar-Geva, M.D. Ph.D., Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology. The Istanbul consensus workshop on embryo assessment: proceedings of an expert meeting. Hum Reprod. 2011 Jun;26(6):1270-83. doi: 10.1093/humrep/der037. Epub 2011 Apr 18. PMID 21502182
- [Background] Kirkegaard K, Ahlstrom A, Ingerslev HJ, Hardarson T. Choosing the best embryo by time lapse versus standard morphology. Fertil Steril. 2015 Feb;103(2):323-32. doi: 10.1016/j.fertnstert.2014.11.003. Epub 2014 Dec 17. PMID 25527231
- [Background] Practice Committee of the American Society for Reproductive Medicine and the Practice Committee of the Society for Assisted Reproductive Technology. Criteria for number of embryos to transfer: a committee opinion. Fertil Steril. 2013 Jan;99(1):44-46. doi: 10.1016/j.fertnstert.2012.09.038. Epub 2012 Oct 22. PMID 23095140
- [Background] Swain JE. Decisions for the IVF laboratory: comparative analysis of embryo culture incubators. Reprod Biomed Online. 2014 May;28(5):535-47. doi: 10.1016/j.rbmo.2014.01.004. Epub 2014 Jan 27. PMID 24656561
- [Background] Fujiwara M, Takahashi K, Izuno M, Duan YR, Kazono M, Kimura F, Noda Y. Effect of micro-environment maintenance on embryo culture after in-vitro fertilization: comparison of top-load mini incubator and conventional front-load incubator. J Assist Reprod Genet. 2007 Jan;24(1):5-9. doi: 10.1007/s10815-006-9088-3. Epub 2006 Dec 13. PMID 17160731
- [Background] Zhang JQ, Li XL, Peng Y, Guo X, Heng BC, Tong GQ. Reduction in exposure of human embryos outside the incubator enhances embryo quality and blastulation rate. Reprod Biomed Online. 2010 Apr;20(4):510-5. doi: 10.1016/j.rbmo.2009.12.027. Epub 2009 Dec 28. PMID 20129824
- [Background] Armstrong S, Arroll N, Cree LM, Jordan V, Farquhar C. Time-lapse systems for embryo incubation and assessment in assisted reproduction. Cochrane Database Syst Rev. 2015 Feb 27;(2):CD011320. doi: 10.1002/14651858.CD011320.pub2. PMID 25721906
- [Background] Meseguer M, Herrero J, Tejera A, Hilligsoe KM, Ramsing NB, Remohi J. The use of morphokinetics as a predictor of embryo implantation. Hum Reprod. 2011 Oct;26(10):2658-71. doi: 10.1093/humrep/der256. Epub 2011 Aug 9. PMID 21828117
- [Background] Lemmen JG, Agerholm I, Ziebe S. Kinetic markers of human embryo quality using time-lapse recordings of IVF/ICSI-fertilized oocytes. Reprod Biomed Online. 2008 Sep;17(3):385-91. doi: 10.1016/s1472-6483(10)60222-2. PMID 18765009
- [Background] Meseguer M, Rubio I, Cruz M, Basile N, Marcos J, Requena A. Embryo incubation and selection in a time-lapse monitoring system improves pregnancy outcome compared with a standard incubator: a retrospective cohort study. Fertil Steril. 2012 Dec;98(6):1481-9.e10. doi: 10.1016/j.fertnstert.2012.08.016. Epub 2012 Sep 10. PMID 22975113
- [Background] Wong CC, Loewke KE, Bossert NL, Behr B, De Jonge CJ, Baer TM, Reijo Pera RA. Non-invasive imaging of human embryos before embryonic genome activation predicts development to the blastocyst stage. Nat Biotechnol. 2010 Oct;28(10):1115-21. doi: 10.1038/nbt.1686. Epub 2010 Oct 3. PMID 20890283
- [Background] Dal Canto M, Coticchio G, Mignini Renzini M, De Ponti E, Novara PV, Brambillasca F, Comi R, Fadini R. Cleavage kinetics analysis of human embryos predicts development to blastocyst and implantation. Reprod Biomed Online. 2012 Nov;25(5):474-80. doi: 10.1016/j.rbmo.2012.07.016. Epub 2012 Aug 2. PMID 22995750
- [Background] Cruz M, Garrido N, Herrero J, Perez-Cano I, Munoz M, Meseguer M. Timing of cell division in human cleavage-stage embryos is linked with blastocyst formation and quality. Reprod Biomed Online. 2012 Oct;25(4):371-81. doi: 10.1016/j.rbmo.2012.06.017. Epub 2012 Jul 7. PMID 22877944
- [Background] Hlinka D, Kalatova B, Uhrinova I, Dolinska S, Rutarova J, Rezacova J, Lazarovska S, Dudas M. Time-lapse cleavage rating predicts human embryo viability. Physiol Res. 2012;61(5):513-25. doi: 10.33549/physiolres.932287. Epub 2012 Aug 8. PMID 22881225
- [Background] Rubio I, Kuhlmann R, Agerholm I, Kirk J, Herrero J, Escriba MJ, Bellver J, Meseguer M. Limited implantation success of direct-cleaved human zygotes: a time-lapse study. Fertil Steril. 2012 Dec;98(6):1458-63. doi: 10.1016/j.fertnstert.2012.07.1135. Epub 2012 Aug 25. PMID 22925687
- [Background] Azzarello A, Hoest T, Mikkelsen AL. The impact of pronuclei morphology and dynamicity on live birth outcome after time-lapse culture. Hum Reprod. 2012 Sep;27(9):2649-57. doi: 10.1093/humrep/des210. Epub 2012 Jun 26. PMID 22740496
- [Background] Aguilar J, Motato Y, Escriba MJ, Ojeda M, Munoz E, Meseguer M. The human first cell cycle: impact on implantation. Reprod Biomed Online. 2014 Apr;28(4):475-84. doi: 10.1016/j.rbmo.2013.11.014. Epub 2013 Dec 11. PMID 24581982
- [Background] Hashimoto S, Kato N, Saeki K, Morimoto Y. Selection of high-potential embryos by culture in poly(dimethylsiloxane) microwells and time-lapse imaging. Fertil Steril. 2012 Feb;97(2):332-7. doi: 10.1016/j.fertnstert.2011.11.042. Epub 2012 Jan 2. PMID 22217963
- [Background] Conaghan J, Chen AA, Willman SP, Ivani K, Chenette PE, Boostanfar R, Baker VL, Adamson GD, Abusief ME, Gvakharia M, Loewke KE, Shen S. Improving embryo selection using a computer-automated time-lapse image analysis test plus day 3 morphology: results from a prospective multicenter trial. Fertil Steril. 2013 Aug;100(2):412-9.e5. doi: 10.1016/j.fertnstert.2013.04.021. Epub 2013 May 28. PMID 23721712
- [Background] VerMilyea MD, Tan L, Anthony JT, Conaghan J, Ivani K, Gvakharia M, Boostanfar R, Baker VL, Suraj V, Chen AA, Mainigi M, Coutifaris C, Shen S. Computer-automated time-lapse analysis results correlate with embryo implantation and clinical pregnancy: a blinded, multi-centre study. Reprod Biomed Online. 2014 Dec;29(6):729-36. doi: 10.1016/j.rbmo.2014.09.005. Epub 2014 Sep 21. PMID 25444507
- [Background] Rubio I, Galan A, Larreategui Z, Ayerdi F, Bellver J, Herrero J, Meseguer M. Clinical validation of embryo culture and selection by morphokinetic analysis: a randomized, controlled trial of the EmbryoScope. Fertil Steril. 2014 Nov;102(5):1287-1294.e5. doi: 10.1016/j.fertnstert.2014.07.738. Epub 2014 Sep 11. PMID 25217875
- [Background] Yang Z, Zhang J, Salem SA, Liu X, Kuang Y, Salem RD, Liu J. Selection of competent blastocysts for transfer by combining time-lapse monitoring and array CGH testing for patients undergoing preimplantation genetic screening: a prospective study with sibling oocytes. BMC Med Genomics. 2014 Jun 22;7:38. doi: 10.1186/1755-8794-7-38. PMID 24954518
- [Background] Morbeck DE, Krisher RL, Herrick JR, Baumann NA, Matern D, Moyer T. Composition of commercial media used for human embryo culture. Fertil Steril. 2014 Sep;102(3):759-766.e9. doi: 10.1016/j.fertnstert.2014.05.043. Epub 2014 Jul 4. PMID 24998366
- [Background] Basile N, Morbeck D, Garcia-Velasco J, Bronet F, Meseguer M. Type of culture media does not affect embryo kinetics: a time-lapse analysis of sibling oocytes. Hum Reprod. 2013 Mar;28(3):634-41. doi: 10.1093/humrep/des462. Epub 2013 Jan 12. PMID 23315059
- [Background] Ciray HN, Aksoy T, Goktas C, Ozturk B, Bahceci M. Time-lapse evaluation of human embryo development in single versus sequential culture media--a sibling oocyte study. J Assist Reprod Genet. 2012 Sep;29(9):891-900. doi: 10.1007/s10815-012-9818-7. Epub 2012 Jun 20. PMID 22714134
- [Background] Goodman LR, Goldberg J, Falcone T, Austin C, Desai N. Does the addition of time-lapse morphokinetics in the selection of embryos for transfer improve pregnancy rates? A randomized controlled trial. Fertil Steril. 2016 Feb;105(2):275-85.e10. doi: 10.1016/j.fertnstert.2015.10.013. Epub 2015 Oct 29. PMID 26522611